CLINICAL TRIAL: NCT03000907
Title: Efficacy of a Multimodal Intervention in the Prevention of Frailty in Obese Elderly People and Study of the Pathophysiological Mechanisms Involved
Brief Title: Efficacy of an Intervention to Prevent Frailty in Obese Elderly People (PRE-FROB)
Acronym: PRE-FROB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 60/16
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Fragility; Sarcopenia; Obese; Elderly
Keywords: prevention; frailty; obese; elderly; physical exercise
MeSH Terms: conditions — Sarcopenia; Obesity; Frailty; Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): * diet: assessment of nutritional status and nutritional requirements and establishment of personalized nutritional plan with monthly dietetic controls.
  * physical exercise: a multi-component physical exercise program that will include aerobic exercise and strengthening, balance and flexibility exercises as well as a weekly group session of health education, during six months.
  Interventions: Other: Intervention
- Control (No Intervention): Clinical practise

INTERVENTIONS:
Other: Intervention — Diet and physical exercises
  Arms: Intervention

SUMMARY:
Rationale: There is increasing evidence that obesity may be a risk factor for frailty in the elderly. Obesity favors a state of chronic inflammation and insulin resistance, involves a fatty infiltration of the muscle and an increased cardiovascular risk and, in addition, obese people usually perform less physical activity. All this favors the loss of mass and muscular function (sarcopenia), a key component of the fragility and the functional deterioration.

Objectives: To evaluate the effectiveness of a multimodal intervention to lose weight in the prevention of frailty in obese elderly people, as well as to know the main mechanisms involved in the frailty process.

Methodology: Design: Controlled, randomized, open-label clinical trial with two parallel intervention arms and 2 years follow-up. Study population: People between 65 and 75 years of age, obese (BMI ≥30), without criteria of fragility and living in the community. Study intervention: multimodal and personalized intervention with the support of a "personal trainer" that has two main axes of action: a) diet: assessment of nutritional status and nutritional requirements and establishment of personalized nutritional plan with monthly dietetic controls and b) physical exercise: a multi-component physical exercise program that will include aerobic exercise and strengthening, balance and flexibility exercises as well as a weekly group session of health education, during six months. Main outcome measures (to be evaluated annually for 2 years): Fragility (according to the L Fried criteria) and Sarcopenia (according to the criteria of the European Working Group on Sarcopenia in Older People -EWGSOP). Sarcopenia is considered if there is a decrease in gait velocity or muscle grip strength (measured with a dynamometer) and a decrease in muscle mass assessed by bioimpedance (BIA). Intermediate outcome measures (at 6, 12 and 24 months): a) weight loss, b) changes in body composition and distribution of body fat, c) glycemic control (HbA1) and insulin resistance (by HOMA index (HOmeostasis Model Assessment)), d) cardiovascular risk according to the REGICOR algorithm, e) functional capacity (according to Barthel Index and 2 Minute Walking Test), f) inflammatory markers (IL-6, CRP(C reactive protein), TNF(Tumor Necrosis Factor)-alpha and leptin) and g) anabolic hormones (IGF-1, ghrelin and testosterone).

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30 and 39 kg / m2
* Non Frail according to L. Fried criteria
* At least one of the following diagnoses:

  * Oral glucose intolerance or type 2 diabetes without insulin therapy.
  * Dyslipidemia (cholesterolemia> 200 mg / dl or triglyceridemia> 150 mg / dl)
  * Arterial hypertension (AT> 120/90 mm Hg)
  * Relevant physical limitations due to obesity
  * Sleep apnea-hypopnea syndrome (SAHS)
* Give written informed consent to participate in the study.

Exclusion Criteria:

* Dementia or other neurodegenerative diseases (Parkinson's disease)
* Neuromuscular diseases
* Severe psychiatric illness that, at the discretion of the physician, prevents good compliance with the study intervention
* Active cancer
* Life expectancy less than 6 months
* Hemiplegia secondary to stroke
* Amputation of a member
* Bariatric surgery tributary patient
* Institutionalized patient

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 319 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Frailty | two years
  Frailty by L Fried criteria

SECONDARY OUTCOMES:
Sarcopenia | two years
  Sarcopenia by European Working Group on Sarcopenia in Older People criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari del Maresme, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No